CLINICAL TRIAL: NCT06336057
Title: Mentalizating in Adults Suffering from Narcolepsy Type 1, a Comparative Prospective Study.
Brief Title: Mentalizating in Adults Suffering from Narcolepsy Type 1.
Acronym: NARCOMENTAL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0408
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Narcolepsy Type 1
Keywords: Narcolepsy type 1; Mentalization; Reflective functioning questionnaire; Mental states task
MeSH Terms: interventions — Mentalization-Based Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Group of patients with narcolepsy type 1.
  Interventions: Behavioral: Mentalization
- Controls: Group of control patients with Obstructive Sleep Apnea (OSA) corrected by treatments
  Interventions: Behavioral: Mentalization

INTERVENTIONS:
Behavioral: Mentalization — complete several questionnaires including the RFQ (reflective functioning questionnaire) and the MST (Mental states task) which are validated questionnaires about mentalization

SUMMARY:
The main objective is to examine the potential mentalization impairments affecting a population suffering from narcolepsy type 1. Indeed, the hypothesis of this research is that mentalization could be impaired in narcoleptic patients.

DETAILED DESCRIPTION:
Narcolepsy type 1 (NT1) is a rare and still poorly understood pathology which can have a significant impact on patient's daily life. Beyond the experience of their chronic illness, their feelings about the difficulties they go through during their lives seem relatively blunted, as if what could be described as restrictive could be acceptable for them. Moreover, the response generated by constraint, even if it is a refusal, rarely turns out to be impulsive or aggressive.

Rapid Eye Movement (REM) sleep is known to play a role in emotional regulation and also in narcolepsy. These processes both take place in hypothalamus, so, a link between them seems conceivable. Surprisingly, the studies about depression, impulsivity, addictions, facial emotional recognition in narcoleptic patients show results that differs from the expectations of the investigators, and can even be at the opposite. It appears difficult to have a clear idea of the mental state of narcoleptic patients.

Mentalization is a concept with a strong empirical base. It corresponds to ability to understand the mental state, of oneself or others, that underlies overt behaviour. The idea of this research is that this process is modified in narcoleptic patients.

The main objective is to examine the potential mentalization impairments affecting a population suffering from narcolepsy type 1. To realise this study a group of patients with NT1 and a control group will complete several questionnaires which are validated about mentalization and other ones. This combination of questionnaire is designed to evaluate the comparability of the groups and search for potential confounding factors.

ELIGIBILITY:
Inclusion Criteria:

For the NT1 patient group:

* Adult patient having been diagnosed with type 1 narcolepsy according to ICSD 3 criteria and the completion of a 48-hour polysomnography at the Sleep Laboratory
* Patient affiliated to or beneficiary of a social security system

For the control group:

* Patient over 18 years old
* Patient followed at Toulouse University Hospital and treated for Obstructive sleep apnea (OSA) with a residual AHI <5/h, demonstrating the absence of residual OSA under treatment
* Patient affiliated to or beneficiary of a social security system

Exclusion Criteria:

* Patient with a history of autism spectrum disorder, chronic psychotic disorder, or bipolar disorder.
* Patient with a history of cognitive disorders of neurological origin
* Patient with a linguistic level in French that does not allow sufficient understanding to complete the questionnaires
* Patient under legal protection measure, under guardianship or curatorship
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients recruited are patients currently followed in the Narcolepsy and Rare Hypersomnia Competence Center at Toulouse University Hospital, with a diagnosis of NT1.
  The witnesses are people followed in the sleep unit of the Toulouse University Hospital in the context of treated OSA.
  All participants will be contacted by telephone or during a follow-up consultation to ask them to participate in this study. An information sheet will be provided to them by mail or in person.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of mentalization abilities, in a population of patients with NT1 versus a control group. | During the inclusion visit
  Scores obtained for the two sub-dimensions of the Reflective functioning questionnaire (RFQ) scale: RFQc and RFQu

SECONDARY OUTCOMES:
Comparison and description of mentalization abilities in a population of patients versus controls. | During the inclusion visit
  comparison of Mental states task scale
Better characterization of the clinical impression of an altered subjective experience of the difficulties the patients are going through. | During the inclusion visit
  comparison of Satisfaction with life scale
Determination of the existence of a correlation between the time of appearance of the first symptoms and the initiation of treatment and the level of mentalization in NT1 patients, or not. | During the inclusion visit
  Time between the appearance of the first symptoms of narcolepsy and the initiation of treatment (only in the patient group)
Determination of the existence of a correlation between the age at the first symptoms of NT1 patients and mentalization abilities, or not. | During the inclusion visit
  Age at the first symptoms of narcolepsy (only in the patient group)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel DEBS, MD, Principal Investigator — Centre de compétence Narcolepsies et Hypersomnies rares, CHU de Toulouse, Hôpital Pierre-Paul Riquet
Locations (1):
- University Hospital Toulouse, Centre de compétence Narcolepsies et Hypersomnies rares, Hôpital Pierre-Paul Riquet, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barateau L, Jaussent I, Lopez R, Boutrel B, Leu-Semenescu S, Arnulf I, Dauvilliers Y. Smoking, Alcohol, Drug Use, Abuse and Dependence in Narcolepsy and Idiopathic Hypersomnia: A Case-Control Study. Sleep. 2016 Mar 1;39(3):573-80. doi: 10.5665/sleep.5530. PMID 26564129
- [Background] Barateau L, Liblau R, Peyron C, Dauvilliers Y. Narcolepsy Type 1 as an Autoimmune Disorder: Evidence, and Implications for Pharmacological Treatment. CNS Drugs. 2017 Oct;31(10):821-834. doi: 10.1007/s40263-017-0464-6. PMID 28940143
- [Background] Bayard S, Abril B, Yu H, Scholz S, Carlander B, Dauvilliers Y. Decision making in narcolepsy with cataplexy. Sleep. 2011 Jan 1;34(1):99-104. doi: 10.1093/sleep/34.1.99. PMID 21203380
- [Background] Beaulieu-Pelletier G, Bouchard MA, Philippe FL. Mental States Task (MST): development, validation, and correlates of a self-report measure of mentalization. J Clin Psychol. 2013 Jul;69(7):671-95. doi: 10.1002/jclp.21942. Epub 2012 Dec 20. PMID 23280811
- [Background] Fonagy P, Luyten P, Moulton-Perkins A, Lee YW, Warren F, Howard S, Ghinai R, Fearon P, Lowyck B. Development and Validation of a Self-Report Measure of Mentalizing: The Reflective Functioning Questionnaire. PLoS One. 2016 Jul 8;11(7):e0158678. doi: 10.1371/journal.pone.0158678. eCollection 2016. PMID 27392018
- [Background] Li X, Sanford LD, Zong Q, Zhang Y, Tan L, Li T, Ren R, Zhou J, Han F, Tang X. Prevalence of Depression or Depressive Symptoms in Patients with Narcolepsy: a Systematic Review and Meta-Analysis. Neuropsychol Rev. 2021 Mar;31(1):89-102. doi: 10.1007/s11065-020-09443-7. Epub 2020 Jul 15. PMID 32671534
- [Background] Luyten P, Campbell C, Allison E, Fonagy P. The Mentalizing Approach to Psychopathology: State of the Art and Future Directions. Annu Rev Clin Psychol. 2020 May 7;16:297-325. doi: 10.1146/annurev-clinpsy-071919-015355. Epub 2020 Feb 5. PMID 32023093
- [Background] Muller S, Wendt LP, Spitzer C, Masuhr O, Back SN, Zimmermann J. A Critical Evaluation of the Reflective Functioning Questionnaire (RFQ). J Pers Assess. 2022 Sep-Oct;104(5):613-627. doi: 10.1080/00223891.2021.1981346. Epub 2021 Oct 1. PMID 34597256
- [Background] Perroud N, Badoud D, Weibel S, Nicastro R, Hasler R, Kung AL, Luyten P, Fonagy P, Dayer A, Aubry JM, Prada P, Debbane M. Mentalization in adults with attention deficit hyperactivity disorder: Comparison with controls and patients with borderline personality disorder. Psychiatry Res. 2017 Oct;256:334-341. doi: 10.1016/j.psychres.2017.06.087. Epub 2017 Jun 30. PMID 28675858
- [Background] Pessoa L. A Network Model of the Emotional Brain. Trends Cogn Sci. 2017 May;21(5):357-371. doi: 10.1016/j.tics.2017.03.002. Epub 2017 Mar 28. PMID 28363681
- [Background] Tohme P, Grey I, Abi-Habib R. The Mental States Task (MST): Correlates and New Perspectives on Mentalizing in a Lebanese Student Sample. J Pers Assess. 2021 Jul-Aug;103(4):498-508. doi: 10.1080/00223891.2020.1769114. Epub 2020 Jun 4. PMID 32496883
- See also: Dauvilliers, Yves. " PNDS narcolepsie type 1 et 2 ". HAS, s. d. — https://www.has-sante.fr/upload/docs/application/pdf/2021-10/texte_pnds_narcolepsies_annexes.pdf